CLINICAL TRIAL: NCT05192070
Title: Investigation of the Acute Effects of Percussive Massage Treatment and Stretching Exercise on Balance and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bmenek.
Record Dates: First submitted 2021-12-30; First posted 2022-01-14 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Sports Physical Therapy
Keywords: percussion massage therapy; dynamic stretching; static stretching

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know which groups they belongs to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Percussive Massage Group (Experimental): Quadriceps, hamstring and gastrocnemius muscles of the participants will done massage for 3 minutes with a hypervolt massage device.
  Interventions: Other: Percussive Massage Group
- Dynamic stretching group (Experimental): Dynamic stretching will be performed for the quadriceps, hamstring and gastrocnemius muscles of the participants with 10 repetitions.
  Interventions: Other: Dynamic stretching group
- Static stretching group (Experimental): Static stretching will be performed for the quadriceps, hamstring and gastrocnemius muscles of the participants with 10 repetitions.
  Interventions: Other: Static stretching group

INTERVENTIONS:
Other: Percussive Massage Group — Quadriceps, hamstring and gastrocnemius muscles of the participants will done massage for 3 minutes with a hypervolt massage device.
  Arms: Percussive Massage Group
Other: Dynamic stretching group — Dynamic stretching will be performed for the quadriceps, hamstring and gastrocnemius muscles of the participants with 10 repetitions.
  Arms: Dynamic stretching group
Other: Static stretching group — Static stretching will be performed for the quadriceps, hamstring and gastrocnemius muscles of the participants with 10 repetitions.
  Arms: Static stretching group

SUMMARY:
In this study, it was aimed to investigate the acute effects of Percussion Massage Therapy and stretching exercises on balance, horizontal jumping and performance in healthy individuals. It was planned to include 45 individuals in the study. Participants will be randomly divided into 3 groups. Horizontal jumping distance, T-Drill test and balance assessment will be done for all participants. After the evaluation, percussion massage therapy will be given to the 1st group, dynamic stretching exercises to the 2nd group, and static stretching exercises to the 3rd group. All measurements will be repeated after the intervention.

DETAILED DESCRIPTION:
48 healthy individuals meeting the inclusion criteria of Istanbul Medipol University will be included in the study. Individuals who are at a level to perform performance tests, who have not undergone orthopedic surgery in any of their regions, who do not have problems in running and during sudden turns, and who do not have a professional sports background will be included in the study. Individuals with a history of trauma, anatomical deformities and skeletal system fractures, diagnosed orthopedic or rheumatological diseases, being included in the physiotherapy program in the last 6 months, and those with pain in any region will be excluded from the study. Before the study, demographic information, horizontal jump test, T-Test and Fizyosoft balance system will be evaluated with both feet and one foot with eyes open and closed. After the evaluation, percussion massage therapy will be given to the 1st group, dynamic stretching exercises to the 2nd group, and static stretching exercises to the 3rd group. All measurements will be repeated after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Capable of performing performance tests
* Those who have not undergone orthopedic surgery in any region
* Having no problems during running and sudden turns
* Individuals who do not have a professional sports background

Exclusion Criteria:

* Trauma history
* Anatomical deformities and skeletal system fractures
* Diagnosed orthopedic or rheumatological diseases
* Being included in a physiotherapy program in the last 6 months
* Individuals with pain in any part of the study

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Horizontal jumping test | 2 minutes
  The starting line is drawn on a flat surface. A tape measure is placed on the floor from the starting line forward and the athletes are asked to take a position with the tips of both toes pointing towards the back of the previously determined line. The distance jumped is measured in cm after the athletes are asked to have their knees bent while their arms are parallel to the floor and knees, and to jump forward as much as possible by swinging their arms and legs quickly.
T drills test | 3 minutes
  It consists of a 9.14 meter forward sprint, 4.57 meter side step to the left, 9.14 meter slide step to the right, 4.57 meter side step to the left, and 9.14 meter backward steps. From the starting point, before starting the run, the individuals are told to take a forward bending motion for at least 3 seconds. The results of the measurement are recorded in seconds. The best score in three attempts will be recorded.
BecureBalance measurement | 10 minutes
  Fizyosoft Becure Balance System balance evaluation protocol will be evaluated as 30 seconds of two-foot balance with eyes open and closed, and 30 seconds of balance with one foot with eyes open and closed.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Menek, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will publish the result of this study for sharing the information about the participants with the other researchers.

REFERENCES:
- [Result] Konrad A, Glashuttner C, Reiner MM, Bernsteiner D, Tilp M. The Acute Effects of a Percussive Massage Treatment with a Hypervolt Device on Plantar Flexor Muscles' Range of Motion and Performance. J Sports Sci Med. 2020 Nov 19;19(4):690-694. eCollection 2020 Dec. PMID 33239942
- See also: The Acute Effects of a Percussive Massage Treatment with a Hypervolt Device on Plantar Flexor Muscles' Range of Motion and Performance — https://pubmed.ncbi.nlm.nih.gov/33239942/